CLINICAL TRIAL: NCT06951165
Title: Investigation of the Effects of Parent-Supported Psychosocial Development Program on 1-3 Year-Old Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Havva Kaçan, ASSOCIATE PROFESSOR, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-KAEK-71
Record Dates: First submitted 2025-02-14; First posted 2025-04-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Children; Parent Child Relationships; Psychosocial Development
Keywords: psychosocial development; Parent; children

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parent-Supported Psychosocial Development Program (Experimental): Parent-Supported Psychosocial Development Program. This program aims to support the psychosocial development of parents of children aged 1-3.
  Interventions: Behavioral: Parent Supported Psychosocial Development Programme
- Active Comparator (Active Comparator): Control group the control group will continue to receive routine check-ups.
  Interventions: Behavioral: Parent Supported Psychosocial Development Programme

INTERVENTIONS:
Behavioral: Parent Supported Psychosocial Development Programme — A six-module online program was developed for parents of children ages 1 to 3. The program was provided to parents as a PDF, one module per week, and each module was discussed online.

SUMMARY:
Growth within the periods of 1-3 years of age, children's physical, psychosocial, It has an important place in terms of cognitive and language development. During this period, children can develop They gain very important skills for their development. In this context, the research the aim of the parent-supported psychosocial development programme for 1-3 year olds is to examine the effects on children. The research is a randomised parallel controlled study. The sample of the study consisted of parents with children between the ages of 1-3 years will constitute. In the study, parents were randomised to the intervention (n:41) and control (n:41) groups. Parent-supported psychosocial development programme will be applied to the intervention group. The control group will be will continue their routine childcare. The data will be analysed with data collection tools will be collected at the same time for both groups. Data collection phase at the end of the programme After the end of the programme, all parents from the control group who requested the training were given the programme.

will be applied in the same way.

DETAILED DESCRIPTION:
Growth within the periods of 1-3 years of age, children's physical, psychosocial, It has an important place in terms of cognitive and language development. During this period, children can develop They gain very important skills for their development. In this context, the research the aim of the parent-supported psychosocial development programme for 1-3 year olds is to examine the effects on children. The research is a randomised parallel controlled study. The sample of the study consisted of parents with children between the ages of 1-3 years will constitute. In the study, parents were randomised to the intervention (n:41) and control (n:41) groups. Parent-supported psychosocial development programme will be applied to the intervention group. The control group will be will continue their routine childcare. The data will be analysed with data collection tools will be collected at the same time for both groups. Data collection phase at the end of the programme After the end of the programme, all parents from the control group who requested the training were given the programme.

will be applied in the same way.

ELIGIBILITY:
Inclusion Criteria:

1. Being a parent of a child between the ages of 1-3
2. Having a tablet, computer or smartphone with internet access

Exclusion Criteria:

1. Using psychiatric medication
2. Being a parent of a child diagnosed with any behavioral problem

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
The level of psychosocial support of parents of children with autism will be measured | four week
  The level of psychosocial support of children's parents will be measured with the Psychosocial Status Assessment Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Güven Hospital, Kastamonu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No